CLINICAL TRIAL: NCT05985408
Title: Left Ventricular Septal Pacing Based Rescue CRT Versus Right Ventricular Apical Pacing Based CRT for Chronic Heart Failure: a Randomized Controlled Trial
Brief Title: LVSP Based CRT vs. RVAP Based CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Li Xiaofei, Doctor, Fu Wai Hospital, Beijing, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0801
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure; Cardiac Resynchronization Therapy; Left Ventricular Septal Pacing; Right Ventricular Septal Pacing
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LVSP-CRT (Experimental): Patients received LVSP based CRT implantation; LVSP, left ventricular septal pacing; CRT, cardiac resynchronization therapy.
  Interventions: Device: left ventricular septal pacing
- RVAP-CRT (Active Comparator): Patients received RVAP based CRT implantation; RVAP, right ventricular apical pacing; CRT, cardiac resynchronization therapy.
  Interventions: Device: right ventricular apical pacing

INTERVENTIONS:
Device: left ventricular septal pacing — For left bundle branch pacing (LBBP) failure cases, use left ventricular septal pacing instead of LBBP; others were same as traditional CRT.
  Arms: LVSP-CRT
Device: right ventricular apical pacing — For left bundle branch pacing (LBBP) failure cases, use right ventricular apical pacing instead of LBBP; others were same as traditional CRT.
  Arms: RVAP-CRT

SUMMARY:
To find out whether left ventricular septal pacing (LVSP)-based cardiac resynchronization therapy (CRT) is superior to right ventricular apical pacing (RVAP)-based CRT in patients with failed left bundle branch pacing at the beginning of chronic heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic heart failure, LVEF ≤35% after at least 3 months of guideline-optimized drug therapy, NYHA class II-IV with complete left bundle branch block (QRSd≥130 ms), OR Atrioventricular block with LVEF ≤ 50% with the indication of cardiac pacing; 3. Age between 18 and 90 years old; 4. The expected survival period is greater than 12 months; 5. Signed the informed consent form for the study.

Exclusion Criteria:

1. Previous mechanical tricuspid valve replacement.
2. Previous pacemaker or other devices implanted and for device replacement or upgrading for this time.
3. Patients have a history of unstable angina, acute myocardial infarction, CABG, and PCI surgery within three months.
4. Persistent atrial fibrillation without AV block, the proportion of biventricular pacing is not expected to less than 95%.
5. Patients participated in any of the other studies at the same time, which may confound the results of this study.
6. Pregnancy, planning to become pregnant.

8. Patients with a history of heart transplantation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
left ventricular ejection fraction (LVEF) | 6 months
  LVEF evaluated by echocardiography，Bi-plane Simpson's method
left ventricular ejection fraction (LVEF) | 12 months
  LVEF evaluated by echocardiography，Bi-plane Simpson's method
left ventricular end-systolic volume (LVESV) | 6 months
  LVESV evaluated by echocardiography
left ventricular end-systolic volume (LVESV) | 12 months
  LVESV evaluated by echocardiography

SECONDARY OUTCOMES:
paced QRSd duration. | 6 months
  QRS duration measurement after the procedure
paced QRSd duration. | 12 months
  QRS duration measurement after the procedure
NT-proBNP | 6 months
  Serum NT-proBNP level
NT-proBNP | 12 months
  Serum NT-proBNP level
6-minute hall walk distance | 6 months
  6-minute hall walk distance
6-minute hall walk distance | 12 months
  6-minute hall walk distance
Heart failure rehospitalization | 6 months
  Rehospitalization due to the exacerbation of heart failure
Heart failure rehospitalization | 12 months
  Rehospitalization due to the exacerbation of heart failure
Rehospitalization for cardiovascular adverse events | 12 months
  Rehospitalization for cardiovascular adverse events
Malignant ventricular arrhythmias | 6 months
  ICD therapy for ventricular tachycardia or ventricular fibrillation
Malignant ventricular arrhythmias | 12 months
  ICD therapy for ventricular tachycardia or ventricular fibrillation
All cause death | 6 months
  All cause death events
All cause death | 12 months
  All cause death events

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ferrick AM, Raj SR, Deneke T, Kojodjojo P, Lopez-Cabanillas N, Abe H, Boveda S, Chew DS, Choi JI, Dagres N, Dalal AS, Dechert BE, Frazier-Mills CG, Gilbert O, Han JK, Hewit S, Kneeland C, DeEllen Mirza S, Mittal S, Ricci RP, Runte M, Sinclair S, Alkmim-Teixeira R, Vandenberk B, Varma N. 2023 HRS/EHRA/APHRS/LAHRS expert consensus statement on practical management of the remote device clinic. Heart Rhythm. 2023 Sep;20(9):e92-e144. doi: 10.1016/j.hrthm.2023.03.1525. Epub 2023 May 19. PMID 37211145
- [Result] Zhang J, Zhang Y, Sun Y, Chen M, Wang Z, Ma C. Success rates, challenges and troubleshooting of left bundle branch area pacing as a cardiac resynchronization therapy for treating patients with heart failure. Front Cardiovasc Med. 2023 Jan 10;9:1062372. doi: 10.3389/fcvm.2022.1062372. eCollection 2022. PMID 36704478
- [Result] Curila K, Jurak P, Jastrzebski M, Prinzen F, Waldauf P, Halamek J, Vernooy K, Smisek R, Karch J, Plesinger F, Moskal P, Susankova M, Znojilova L, Heckman L, Viscor I, Vondra V, Leinveber P, Osmancik P. Left bundle branch pacing compared to left ventricular septal myocardial pacing increases interventricular dyssynchrony but accelerates left ventricular lateral wall depolarization. Heart Rhythm. 2021 Aug;18(8):1281-1289. doi: 10.1016/j.hrthm.2021.04.025. Epub 2021 Apr 28. PMID 33930549